CLINICAL TRIAL: NCT04990349
Title: Normoxemic Versus Hyperoxemic Extracorporeal Oxygenation : Impact on Organ Dysfunction in Patients Supported by Veino-arterial ECMO for Cardiogenic Shock
Brief Title: Normoxemic Versus Hyperoxemic Extracorporeal Oxygenation in Patients Supported by Veino-arterial ECMO for Cardiogenic Shock
Acronym: ECMOxy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECMOxy - pilot study
Record Dates: First submitted 2021-07-30; First posted 2021-08-04 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2023-09

CONDITIONS: Cardiogenic Shock; Extracorporeal Membrane Oxygenation
Keywords: Cardiogenic shock; Extracorporeal Membrane Oxygenation; Hyperoxia
MeSH Terms: conditions — Shock, Cardiogenic; Hyperoxia | interventions — nitrox

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal normoxemia (Experimental): * After randomization, extracorporeal normoxemia is targeted by setting the ECMO membrane oxygen fraction (FmO2) at 60%.
  * The objective is to maintain oxygen partial pressure measured on the arterial cannula (PO2 postoxygenator) between 100 and 150 mmHg.
  * PO2 postoxygenator is monitored at least twice a day by the nurse.
  * If PO2 postoxygenator is less than 100 mmHg or more than 150 mmHg, FmO2 is modified by 10% and PO2 postoxygenator is monitored 10 minutes after.
  * Ventilator's setting at let to the clinician's discretion. However, PaO2 on right radial artery will be monitored to ensure that is more that 80 mmHg.
  * Intervention will be applied for 7 days after randomization.
  Interventions: Drug: Oxygen gas
- Extracorporeal hyperoxemia (Active Comparator): * After randomization, extracorporeal hyperoxemia is targeted by setting the ECMO membrane oxygen fraction (FmO2) at 100%.
  * The objective is to maintain PO2 postoxygenator higher than 300 mmHg.
  * PO2 postoxygenator is monitored at least twice a day by the nurse.
  * If PO2 postoxygenator is less than 300 mmHg, membrane change should be discussed.
  * Ventilator's setting at let to the clinician's discretion. However, PaO2 on right radial artery will be monitored to ensure that is more that 80 mmHg.
  * Intervention will be applied for 7 days after randomization.
  Interventions: Drug: Oxygen gas

INTERVENTIONS:
Drug: Oxygen gas — Targeted PO2 postoxygenator is obtained by modulating ECMO Membrane oxygen fraction.

SUMMARY:
Because of dual oxygenation and oxygenator performance (PO2 postoxygenator up to 500 mmHg), hyperoxemia (PaO2 > 150 mmHg) is frequent in veino-arterial ECMO, especially in the lower part of the body, which is mainly oxygenated by ECMO.

By enhancing oxygen free radicals' production, hyperoxemia might favor gut, kidney and liver dysfunction.

We hypothesize that targeting an extracorporeal normoxemia (i.e. PO2 postoxygenator between 100 and 150 mmHg) will decrease gut, kidney and liver dysfunctions, compared to a liberal extracorporeal oxygenation.

DETAILED DESCRIPTION:
Randomization:

Patients will be randomized in the 6 hours following ECMO start in the normoxemia or in the hyperoxemia group. Randomization will be stratified on center, and medical or postcardiotomy indication for ECMO.

Description of experimental arm (Normoxemia group):

* After randomization, extracorporeal normoxemia is targeted by setting the ECMO membrane oxygen fraction (FmO2) at 60%.
* The objective is to maintain oxygen partial pressure measured on the arterial cannula (PO2 postoxygenator) between 100 and 150 mmHg.
* PO2 postoxygenator is monitored at least twice a day by the nurse.
* If PO2 postoxygenator is less than 100 mmHg or more than 150 mmHg, FmO2 is modified by 10% and PO2 postoxygenator is monitored 10 minutes after.
* Ventilator's settings at let to the clinician's discretion. However, PaO2 on right radial artery will be monitored to ensure that is more that 80 mmHg.
* Intervention will be applied for 7 days after randomization.

Description of the control arm (Hyperoxemia group):

* After randomization, extracorporeal hyperoxemia is targeted by setting the ECMO membrane oxygen fraction (FmO2) at 100%.
* The objective is to maintain PO2 postoxygenator higher than 300 mmHg.
* PO2 postoxygenator is monitored at least twice a day by the nurse.
* If PO2 postoxygenator is less than 300 mmHg, membrane change should be discussed.
* Ventilator's setting at let to the clinician's discretion. However, PaO2 on right radial artery will be monitored to ensure that is more that 80 mmHg.
* Intervention will be applied for 7 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patient supported by veino-arterial ECMO for cardiogenic shock for less than 6 hours
* Affiliation to social protection

Exclusion Criteria:

* Age < 18 years old
* Pregnancy
* Opposition of the patient or his relatives
* Cannulation during cardiopulmonary resuscitation
* Cardiopulmonary resuscitation duration > 10 minutes before ECMO implantation
* Patient moribound on the day of randomization
* Chronic hemodialysis
* Chronic intestinal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-09 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Enterocyte damage | At day 2
  Plasma Intestinal Fatty Acid Biding Protein (I-FABP) concentration

SECONDARY OUTCOMES:
Feasibility of the oxygenation protocol | From day 0 to day 6
  Percentage of time in the oxygenation target
Security of the oxygenation protocol | From day 0 to day 6
  Number of right radial PaO2 below 80 mmHg
Organ failure | From day 0 to day 30
  Death or severe stroke (NIHSS > 11) or mesenteric ischemia
Organ failure | At day 0, day 2 and day 6
  Non cardiac component of the Sequential Organ Failure Assessment (SOFA) score
Organ failure | At day 0, day 2 and day 6
  Plasma lactate concentration
Enterocyte damage | At day 0, and day 1
  Plasma Intestinal Fatty Acid Biding Protein (I-FABP) concentration
Enterocyte function | At day 0 and day 2
  Difference between plasma citrulline concentrations at day 0 and day 2
Liver failure | At day 0, day 2 and day 6
  Plasma Aspartate aminotransferase (ASAT) concentration
Liver failure | At day 0, day 2 and day 6
  Prothrombine time
Renal failure | At day 0, day 2 and day 6
  Plasma creatinine concentration
Renal failure | From 0 to day 6
  Need for renal replacement therapy
Systemic inflammation | At day 0, day 2 and day 6
  Plasma CRP, TNF alpha, IL6 and IL8 concentrations
Anti-oxydant stock | At day 0, day 2 and day 6
  Plasma vitamin C, vitamin E, and Glutathion concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: 2023

REFERENCES:
- [Result] Munshi L, Kiss A, Cypel M, Keshavjee S, Ferguson ND, Fan E. Oxygen Thresholds and Mortality During Extracorporeal Life Support in Adult Patients. Crit Care Med. 2017 Dec;45(12):1997-2005. doi: 10.1097/CCM.0000000000002643. PMID 28787294
- [Result] Hayes RA, Shekar K, Fraser JF. Is hyperoxaemia helping or hurting patients during extracorporeal membrane oxygenation? Review of a complex problem. Perfusion. 2013 May;28(3):184-93. doi: 10.1177/0267659112473172. Epub 2013 Jan 15. PMID 23322670
- [Result] Chou HC, Chen CM. Neonatal hyperoxia disrupts the intestinal barrier and impairs intestinal function in rats. Exp Mol Pathol. 2017 Jun;102(3):415-421. doi: 10.1016/j.yexmp.2017.05.006. Epub 2017 May 12. PMID 28506763
- [Result] Falk L, Sallisalmi M, Lindholm JA, Lindfors M, Frenckner B, Broome M, Broman LM. Differential hypoxemia during venoarterial extracorporeal membrane oxygenation. Perfusion. 2019 Apr;34(1_suppl):22-29. doi: 10.1177/0267659119830513. PMID 30966908